CLINICAL TRIAL: NCT05909709
Title: An Open Label Dose Escalation Pilot Study to Evaluate the Safety of Alocyte Delivered Via Intra-articular Facet Injection for the Treatment of Facetogenic Back Pain
Brief Title: Dose Escalation Pilot Study to Evaluate the Safety of Alocyte for the Treatment of Facetogenic Back Pain
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Alimorad Farshchian (Other)
Responsible Party: Sponsor-Investigator, Alimorad Farshchian, Physician Principal Investigator, The Center For Regenerative Medicine Laboratories
Organization: The Center For Regenerative Medicine Laboratories (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 00070133
Record Dates: First submitted 2023-05-25; First posted 2023-06-18 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Facet Joints; Degeneration; Back Pain; Facet Joint Pain
Keywords: Back pain; Facet joint pain
MeSH Terms: conditions — Back Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Alocyte Low dose (Experimental): Subjects will receive low dose injection in a single facet joint
  Interventions: Drug: Alocyte low dose
- Alocyte Medium dose (Experimental): Subjects will receive medium dose injections in three facet joints
  Interventions: Drug: Alocyte medium dose
- Alocyte High dose (Experimental): Subjects will receive high dose injections in five facet joints
  Interventions: Drug: Alocyte high dose

INTERVENTIONS:
Drug: Alocyte low dose — Low dose containing 0.2 - 1.0 x 10^11 particles and 3-10x10^6 cell in 2mL which will be administered intra-facet into a single facet joint.
  Preparation of low dose: 1ml of Alocyte will be diluted with 9ml of saline. After mixing well, only 2ml of the diluted product will be used.
  Arms: Alocyte Low dose
Drug: Alocyte medium dose — Medium dose containing 0.6 - 3.0 x 10^11 particles and 9-30x10^6 cell in 6mL which will be administered intra-facet into three facet joints delivering 2ml/facet joint.
  Preparation of medium dose: 1ml of Alocyte will be diluted with 9ml of saline. After mixing well, only 6ml of the diluted product will be used.
  Arms: Alocyte Medium dose
Drug: Alocyte high dose — High dose containing 1.0 - 5.0 x 10^11 particles and 15-50x10^6 cell in 10mL which will be administered intra-facet into five facet joints delivering 2ml/facet joint.
  Preparation of high dose: 1ml of Alocyte will be diluted with 9ml of saline. After mixing well, 10ml of diluted product will be used.
  Arms: Alocyte High dose

SUMMARY:
The purpose of this study is to see if the use of Alocyte (cord blood plasma plus mononucleic cells) will be safe, well tolerated, and whether it causes any side effects. The study will also examine if the use of the Investigational Product (IP) is able to reduce local inflammation or alleviate Facetogenic back pain

DETAILED DESCRIPTION:
Ghormley, in 1933, was the first to perform oblique spine radiographs to view the zygapophysial or facet joints and coin the term "facet syndrome" to refer to LBP with "sciatica" originating from the facet joints. The facet joint may be affected by systemic disease, such as rheumatoid arthritis and ankylosing spondylitis, or be site of micro traumatic fractures, such as osteoarthritis, meniscoid entrapment, synovial impingement, joint subluxation, synovial inflammation, loss of cartilage, and mechanical injury. Facetogenic pain is the result of repetitive stress and/or cumulative low-level trauma, leading to inflammation and stretching of the joint capsule.

Current treatment options for this disease are limited to symptomatic treatment, including analgesics, physiotherapy, and minimally invasive or surgical treatment (spinal fusion or non-fusion), but none of the methods addresses the underlying problem. The pathological process of intervertebral disc degeneration cannot be prevented by these therapies.

Alocyte is a cellular, minimally manipulated product derived from umbilical cord blood. Alocyte's manufacturing methodology is designed to enrich human umbilical cord plasma and human umbilical cord blood-derived mononuclear cells (hematopoietic lineage cells such as lymphocytes, monocytes, stem and progenitor cells, as well as mesenchymal stem cells) present in full-term cord blood. The final product is composed of a heterogenous population of cellular products, mainly the exosomes, cytokines, and nucleated cells.

Cytokine expression of Alocyte was fully evaluated. Alocyte showed a robust expression of RANTES, Osteopontin, and Angiostatin where the first two are stem cell repair cytokines and the latter is pro-angiogenic cytokine. Other cytokine showed moderate levels are IL-8, PDGF-BB, TIMP-1, TIMP-2, Angiopoietin-1, Angiogenin, MMP-9, Tie-2, uPAR, BDNF, TGF-ß2, GRO, IGFBP-1, IGFBP-2, IL-8, IL-12-p40, MIF, and NAP-2. Alocyte contained a variety of pro-angiogenic, immune-modulatory, anti-inflammatory, pro-metabolism, and tissue repair growth factors.

Therefore, a regenerative approach for treating Facetogenic pain will be beneficial by promoting changes in the pathogenic mechanism triggered by the cellular therapeutic product Alocyte.

ELIGIBILITY:
Inclusion Criteria:

* In order to be eligible to participate in this study, all individuals must meet all of the following criteria:

  1. Subjects age > 18 years at the time of signing the Informed Consent Form.
  2. Male or Female.
  3. Ability of participant to understand and the willingness to sign a written informed consent document.
  4. Facetogenic back pain diagnosed using the following diagnostic criteria Subjects who have chronic low back pain based on clinical evaluation. Pain onset at dorsal extension and release at flexion is often considered suggestive for facet pain, even if non-specific, such as maximal tenderness upon deep palpation of posterior elements.
  5. Patient with up to 5 diseased facet joints
  6. Chronic Facetogenic pain (≥ 6 months) in patients that have failed conservative management
  7. Subjects must be reasonably able to return for multiple follow-up visits.
  8. For Women of Child-Bearing Potential (WOCBP) only, willingness to use FDA-recommended birth control until 6 months post treatment.
  9. Any male subject must agree to use contraceptives and not donate sperm during the study.

Exclusion Criteria:

1. Previous surgical intervention for back pain
2. Previous stem cell injection(s) within the last year
3. Use of anticoagulation or NSAIDs within 5 days of the injection
4. MRI finding of severe high-grade lumbar stenosis
5. Leg pain exceeding back pain
6. Pain worse with flexion maneuvers
7. Fracture of lumbar vertebrae
8. Inability to perform any of the assessments required for endpoint analysis.
9. Clinically significant abnormal screening laboratory or clinical assessment values
10. Use of medications during the early phase of treatment such as chronic narcotic use, systemic corticosteroid administration, local corticosteroid injection at facets anticoagulant therapy and viscosupplementation into facets, any investigational drug used within 3 months prior to screening or during study and surgery in the facets
11. Subjects with serious co-morbidities are excluded.
12. Evidence of inflammatory arthritis (example, rheumatoid arthritis and ankylosing spondylitis) or traumatic fractures, osteoarthritis, meniscoid entrapment, synovial impingement, joint subluxation, synovial inflammation, loss of cartilage, and mechanical injury.
13. Have a clinical history of malignancy within 5 years (i.e., subjects with prior malignancy must be disease free for 5 years), except curatively treated basal cell carcinoma, squamous cell carcinoma, melanoma in situ or cervical carcinoma, if recurrence occurs.
14. Be currently participating (or participated within the previous 6 months) in an investigational therapeutic or device trial.
15. Exhibiting signs of moderate or severe chronic respiratory disease (such as COPD, asthma, or pulmonary fibrosis).
16. Patient with rheumatologic disorders.
17. History of chronic liver disease or patient showing signs of clinical jaundice at the time of screening.
18. History of severe chronic kidney disease or requiring dialysis.
19. Patient with NYHA Class III or IV congestive heart failure or life-threatening arrhythmias.
20. Subjects with a history of bleeding disorders, anticoagulation therapy that cannot be stopped as prior to the treatment.
21. Any unstable condition of clinical significance, e.g., uncontrolled hypertension, unstable angina pectoris, worsening asthma.
22. Hydroxychloroquine, oral or parenteral corticosteroids, immunosuppressants, or immunomodulating agents within 21 days prior to the Day 0/treatment visit.
23. Be a female who is pregnant, nursing, or of childbearing potential while not practicing effective contraceptive methods. Female subjects must undergo a blood pregnancy test at screening which will be within 72 hours of the IP infusion.
24. Subject has a body mass index (BMI) greater than 42 kg/m2
25. Subject has or had an active infection requiring systemic antibiotics within 12 weeks of enrollment in the study
26. Inability to perform any of the assessments required for endpoint analysis.
27. Active listing (or expected future listing) for transplant of any organ.
28. Be a solid organ transplant recipient. This does not include prior cell-based therapy (>12 months prior to enrollment), bone, skin, ligament, tendon or corneal grafting. Have a history of organ or cell transplant rejection.
29. History of drug abuse (illegal "street" drugs except marijuana, if it is legal to use in states where patient resides), or prescription medications not being used appropriately for a pre-existing medical condition or alcohol abuse (≥ 5 drinks/day for ˃ 3 months), or documented medical, occupational, or legal problems arising from the use of alcohol or drugs within the past 24 months
30. Patients with untreated HIV infection. However, patients can be enrolled if have been treated for HIV and the test negative for HIV viral load but still test positive for antibodies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2024-04-29 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Safety of Alocyte treatment adverse events | through study completion, an average of 13 months
  To evaluate safety ( incident of grade 3 or 4 or treatment emergent serious adverse events) of Alocyte administered in subjects experiencing Facetogenic back pain at a low, medium and high dose.
Incidence of treatment emergent adverse events as assessed by complete blood count safety lab tests | at 1 month
  To evaluate the incidence of treatment emergent adverse events as assessed by safety lab blood sample test complete blood count (CBC with differential)
Incidence of treatment emergent adverse events as assessed by complete blood count safety lab tests | at 3 months
  To evaluate the incidence of treatment emergent adverse events as assessed by safety lab blood sample test complete blood count (CBC with differential)
Incidence of treatment emergent adverse events as assessed by complete blood count safety lab tests | at 6 months months
  To evaluate the incidence of treatment emergent adverse events as assessed by safety lab blood sample test complete blood count (CBC with differential)
Incidence of treatment emergent adverse events as assessed by safety complete metabolic panel ab tests | at 1 month
  To evaluate the incidence of treatment emergent adverse events as assessed by safety lab blood sample test complete metabolic panel (CMP)
Incidence of treatment emergent adverse events as assessed by safety complete metabolic panel lab tests | at 3 month
  To evaluate the incidence of treatment emergent adverse events as assessed by safety lab blood sample test complete metabolic panel (CMP)
Incidence of treatment emergent adverse events as assessed by safety complete metabolic panel lab tests | at 6 month
  To evaluate the incidence of treatment emergent adverse events as assessed by safety lab blood sample test complete metabolic panel (CMP)
Incidence of treatment emergent adverse events as assessed by safety coagulation panel lab tests | at 1 month
  To evaluate the incidence of treatment emergent adverse events as assessed by safety lab blood sample test coagulation panel
Incidence of treatment emergent adverse events as assessed by safety coagulation panel lab tests | at 3 months
  To evaluate the incidence of treatment emergent adverse events as assessed by safety lab blood sample test coagulation panel
Incidence of treatment emergent adverse events as assessed by safety coagulation panel lab tests | at 6 months
  To evaluate the incidence of treatment emergent adverse events as assessed by safety lab blood sample test coagulation panel
Incidence of treatment emergent adverse events as assessed by blood biomarker sample lab tests | at 1 month
  To evaluate the incidence of treatment emergent adverse events as assessed by blood biomarker sample test C-reactive protein (CRP)
Incidence of treatment emergent adverse events as assessed by blood biomarker sample lab tests | at 3 months
  To evaluate the incidence of treatment emergent adverse events as assessed by blood biomarker sample test C-reactive protein (CRP)
Incidence of treatment emergent adverse events as assessed by blood biomarker sample lab tests | at 6 months
  To evaluate the incidence of treatment emergent adverse events as assessed by blood biomarker sample test C-reactive protein (CRP)

SECONDARY OUTCOMES:
Efficacy of Alocyte treatment as assessed by the change in Quality of Life (QoL) SF-12 questionnaire | baseline, 1 month, 3 months, 6 months, 12 months
  Change from baseline in subject QoL SF-12 questionnaire consisting of twelve questions that measure eight health domains to assess physical and mental health. Scores range from 0 to 100, with higher scores indicating better physical and mental health functioning
Efficacy of Alocyte Treatment for pain management as assessed by the change in Numeric Rating Scale (NRS) pain scale | baseline, 1 month, 3 months, 6 months, 12 months
  Change between baseline in pain using the Numeric Rating Scale (NRS) on a scale from 0 (equals no pain) to 10 (worst pain imaginable)
Efficacy of Alocyte Treatment for pain as assessed by the change in the Owestry Back Pain questionnaire | baseline, 1 month, 3 months, 6 months, 12 months
  Change between baseline in back pain using Oswestry Low back pain questionnaire made up of 10 questions. Each question is scored from 0-5 (minimum to maximum).

CONTACTS AND LOCATIONS:
Overall Officials: Alimorad Farshchian, MD, Principal Investigator — The Center For Regenerative Medicine Laboratories
Locations (1):
- The Center for Regenerative Medicine, North Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No